CLINICAL TRIAL: NCT07355530
Title: A Randomized Double-blind, Placebo-controlled Trial of Adipose-derived Regenerative Cells Injected Into Corpora Cavernosum Following Radical Prostatectomy
Brief Title: Can Adipose Derived Regenrative Cells be Used for Treating Erectile Dysfunction After Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-005140-33
Record Dates: First submitted 2025-11-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: ED; Adipose Derived Stem Cells

STUDY DESIGN:
Intervention Model Description: performed as a randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): One injection of Ringer Lactate
  Interventions: Other: Placebo
- Active treatment (Experimental): Injection of adipose derived regnerative cells
  Interventions: Drug: Adipose-Derived Regenerative Cells

INTERVENTIONS:
Drug: Adipose-Derived Regenerative Cells — Adipose-derived regenerative cells was injected into the corpus cavernosum.
  Arms: Active treatment
Other: Placebo — Injection of ringer lactate
  Arms: Placebo

SUMMARY:
The goal of this study was to investigate if adipose derived regenerative cells can be used as a treatment for erectile dysfunction following radical prostatectomy.

70 participants were enrolled in the study and was performed as a double- blinded study. 35 participants in the active study arm recieved an injection into the penis of adipose derived regenerative cells, while the participants of the placebo arm recieved a placebo injection.

All 70 participants undervent liposuccion of the abdomen to harvest the adipose derived regenerative cells, and the 35 participants in the active study arm recieved their own regenerative cells.

All participants answered the questionnaires International-Index-of- Erectile function 5 and Erection Hardness Scale before treatment and after 1,3,6 and 12 months. These data was used to evaluate the effect of one injection of adipose derived regenerative cells.

ELIGIBILITY:
Inclusion criteria:

* Nervesparing robot assisted RP
* Erectile dysfunction for more than a year after RP
* Normal erectile function before RP (IIEF-5 > 22) and postoperative IIEF-5 score 5-20 or EHS 1
* Involved in a monogamous, heterosexual relationship (since questionnaires are only valid for heterosexual relationsships), where both parts are interested in sexual activities
* Insufficient effect of standard medical treatment for ED
* Subcutaneous adipose deposits on the abdomen > 120 mL
* Performance status 0
* Ability to give informed consent
* Proficiency in the Danish language to understand the questionnaires IIEF-5 and EHS

Exclusion criteria:

* Problems with general anesthesia
* Incontinence after RP
* Anti-thrombotic treatment that cannot be discontinued or substituted with heparin
* No interest in sexual interaction with a partner
* Previous pelvic surgery or radiation
* Systemic autoimmune disease
* Alcohol or drug abuse

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Changes in International-Index-of-Erectile-Function 5 12 months after intervention | 12 months
  All paticipants answered the questionnaire International-Index-of-Erectile-Function 5 at baseline and after 12 months.
  The questionnaire focus on confidence, erection hardness, maintaining erection and satisfaction during intercourse.
  The scale of the score is from 5 to 25. The higher the score is, the better is the erectile function.
  A score from 5-7 means severe erectile dysfunction A score from 8-11 is moderate erectile dysfunction A score from 12-16 is mild to moderate erectile dysfunction A score from 17-21 is mild erectile dysfunction A score from respresents no erectile dysfunction. A higher score after 12 months means that the erectile function is improved.

SECONDARY OUTCOMES:
Changes in Erectile Hardness Scale (EHS) six months after intervention | 6 months
  Erectile Hardness Scale (EHS) was answered at baseline and 6 months after intervention. The scale are running from 0-4, it is used to rate erection firmness for penetration.
  0: no enlargement at all
  1. Enlarged but not firm
  2. Firm, but not hard enough for penetration
  3. Hard enough for penetration, but not fully rigid
  4. fully rigid and completely hard. A higher score after 6 month means that the erection is better than before intervention.
RigiScan | 6 months
  Changes in RigiScan scores 6 months after intervention. RigiScan is a non- invasive diagnostic devise that are used to measure penile rigidity and circumference changes during sleep. The divice consist of two loops and a monitor, and the loops are able to monitor the erection quality over time, if the values of the data improve 6 months after intervention, is the erection improved.
  We monitored Frequency of erections during sleep (number of erections)
RigiScan data | 6 months
  Changes in RigiScan scores 6 months after intervention. RigiScan is a non- invasive diagnostic devise that are used to measure penile rigidity and circumference changes during sleep. The divice consist of two loops and a monitor, and the loops are able to monitor the erection quality over time, if the values of the data improve 6 months after intervention, is the erection improved.
  We monitored duration of erection during sleep in minutes.
RigiScan data | 6 months
  Changes in RigiScan scores 6 months after intervention. RigiScan is a non- invasive diagnostic devise that are used to measure penile rigidity and circumference changes during sleep. The divice consist of two loops and a monitor, and the loops are able to monitor the erection quality over time, if the values of the data improve 6 months after intervention, is the erection improved.
  We monitored tumescence of erection, the expansion of the circumference in cm.
RigiScan data | 6 months
  Changes in RigiScan scores 6 months after intervention. RigiScan is a non- invasive diagnostic devise that are used to measure penile rigidity and circumference changes during sleep. The divice consist of two loops and a monitor, and the loops are able to monitor the erection quality over time, if the values of the data improve 6 months after intervention, is the erection improved.
  We monitored hardness of erection in %

CONTACTS AND LOCATIONS:
Locations (1):
- Odense Universityhospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data are stored in 'REDCap' that is government approved for storage of personal data, and is used to keep track of the clinical trial data via the Odense Patient data Explorative Network 'OPEN'. The aforementioned questionnaires regarding the erectile function will be filed out by the patients themselves directly into the REDCap patient file via a link.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 of January 2018 til 31 of December 2028
Access Criteria: Sponsor and primary investigator will be able to access the database. Primary investigator can make permission to access the database by creating a login.
  The GCP (good clinical practice) Units investigators can also access the database.
URL: https://open.rsyd.dk/